CLINICAL TRIAL: NCT02002871
Title: Monocenter, Randomized, Intraindividual, Open Label, Exploratory Study Comparing 4 Weeks of Treatment With 453nm Blue Light With no Treatment in Patients With Eczema
Brief Title: Blue Light for Treating Eczema
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Philips Electronics Nederland BV (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EczemaCT01; CIV-13-08-011581 (Other: Unique identification number EUDAMED)
Record Dates: First submitted 2013-12-02; First posted 2013-12-06 (Estimated); Results first posted 2015-07-20 (Estimated); Last update posted 2015-07-20 (Estimated); Status verified 2015-06

CONDITIONS: Eczema
MeSH Terms: conditions — Eczema

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Blue light (Experimental): Irradiation with PSOCT02 device emitting blue light at a wavelength of 453nm
  Interventions: Device: PSO-CT02 device
- Control (No Intervention): contralateral untreated control plaque on the same patient.

INTERVENTIONS:
Device: PSO-CT02 device — The PSO-CT02 device is worn on the affected skin area where it irradiates the target Eczema area for 30 minutes with blue light. A contralateral eczema area is left untreated and serves as control.
  Arms: Blue light

SUMMARY:
Monocenter, randomized, intraindividual, open label, exploratory study comparing 4 weeks of treatment with 453nm blue light with no treatment in patients with Eczema. Patients will be screened up to 28 days before start of treatment. During the screening visit, the purpose and procedures of the study will be explained to potential patients and informed consent will be obtained. In addition, fungal superinfection of the target area will be examined using direct preparations and mycology cultures. At the baseline visit, patients with Eczema will be determined and all inclusion and exclusion criteria will be assessed. For eligible patients, two comparable treatment areas will be randomized to treatment with blue light (target area) or to serve as untreated control area. After randomization, patients will receive treatment of the target area with 3 applications per week at the investigational site for a total treatment period of 4 weeks. During those 4 weeks, safety and effectiveness assessments will be performed at weekly intervals. After end of treatment, the patients will be followed-up for another 2 weeks. In case no full resolution of adverse events occurred at the 2 week follow-up visit, a follow-up call will be performed after another 2 weeks. Treatment responses will be photo documented

ELIGIBILITY:
Inclusion Criteria:

1. Signed and dated informed consent prior to any study-mandated procedure
2. Good health as determined by the Investigator according to physical examination
3. Willing and able to comply with study requirements
4. Skin type I-IV according to Fitzpatrick
5. Eczema, severity defined by an Eczema Area Severity Index (EASI)smaller/equal 20
6. Comparable clinical symptomatology of both intended treatment Areas

8. Reliable method of contraception for women of childbearing potential (i.e. low failure rate less than 1% per year; e.g. oral contraceptives, intrauterine device [IUD] or transdermal contraceptive patch) 9. Willing to abstain from excessive sun / UV exposure (e.g. sunbathe, solarium) during the course of the study

Exclusion Criteria:

1. Inmates of psychiatric wards, prisons, or other state institutions
2. Investigator or any other team member involved in the conduct of the clinical study
3. Participation in another clinical trial within the last 30 days
4. Pregnant and lactating women
5. Photodermatosis and/or Photosensitivity
6. Porphyria and/or hypersensitivity to porphyrins
7. Congenital or acquired immunodeficiency
8. Patients with any of the following conditions present on the study areas; Malignoma of the skin or severe actinic damage of the skin, atypical naevi or signs of hyperpigmentation, precancerosis viral (e.g. herpes or varicella) lesions of the skin, fungal and bacterial skin infections, parasitic infections and atrophic skin
9. Patients with genetic deficiencies attached with increased sensitivity to light or increased risk to dermatologic cancer (i.e. Xeroderma pigmentosum, Cockayne Syndrome, Bloom- Syndrome)
10. Current diagnosis of exfoliative or toxic dermatitis.
11. Evidence of superinfection of the intended treatment areas

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2013-10; Primary Completion 2014-03 (Actual); Study Completion 2014-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Verena von Felbert, PD Dr., Principal Investigator — Klinik for Dermatology and Allergy, medical faculty of the RWTH Aachen
Locations (1):
- Klinik for Dermatology and Allergology, medical faculty of the RWTH Aachen, Aachen, North Rhine-Westphalia, Germany

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Date of first enrollment: 23.10.2013, University Clinic Aachen Date of LPLV: 17.02.2014
Groups:
- Blue Light vs Control: Light wavelength 453nm, compared to contralateral untreated control plaque on the same patient.
  PSO-CT02 device: The PSO-CT02 device is worn on the affected skin area where it irradiates the target Eczema area for 30 minutes with blue light. A contralateral eczema area is left untreated and serves as control.
Period: Overall Study
Arm/Group | Blue Light vs Control
Started | 21
Completed | 20
Not Completed | 1

BASELINE CHARACTERISTICS:
Arm/Group | Blue Light vs Control
Number analyzed (Participants) | 21
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 21
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11
  Male | 10
Region of Enrollment [Number; unit: participants]
  Germany | 21

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline (Visit 2) of the Sum Score of Local Eczema Rating of the Target Area as Compared to the Control Area at End of Treatment
Description: The investigator rated the key symptoms erythema, induration/papulation/edema, excoriation, lichenification and crusts on a score of 0-3 (none, mild, moderate, and severe) with half steps allowed. A total severity score was calculated as the sum of the single symptom ratings (range 0-15 whereas 0 (best) - 15 (worst)).
Time Frame: at week 4
Population: Overall number of participants is also 20 because control and treated plaque were anaylsed on the same patient.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Blue Light: Light wavelength 453nm
  PSO-CT02 device: The PSO-CT02 device is worn on the affected skin area where it irradiates the target Eczema area for 30 minutes with blue light.
Arm/Group | Blue Light | Control
Number analyzed (Participants) | 20 | 20
units on a scale | -1.9 (2.02) | -1.3 (2.24)
Statistical Analysis 1: Comparison: Blue Light vs Control; The statistical analysis was performed on the difference of the change from baseline of the Blue light treated plaque versus the Control plaque; Test type: Superiority or Other; p = 0.0152, t-test, 2 sided

2. Secondary Outcome: Change From Week 4 of the Sum Score of Local Eczema Rating as Compared to the Control Area at End of Follow-up
Description: as for outcome 1
Time Frame: week 6
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Blue Light | Control
Number analyzed (Participants) | 20 | 20
units on a scale | -0.5 (1.54) | -0.5 (1.43)

3. Secondary Outcome: Change From Baseline of Inflammation (Erythema) Evaluated by Mexameter of the Target Area as Compared to the Control Area
Description: Higher values describe higher erythema levels.
Time Frame: week 4, 6
Measure: Mean (Standard Deviation); unit: arbitrary units
Arm/Group | Blue Light | Control
Number analyzed (Participants) | 20 | 20
arbitrary units
  week 4 | 4.7 (8.11) | -0.9 (10.28)
  week 6 | 1.1 (7.74) | 0.3 (7.36)

4. Secondary Outcome: Change From Week 4 (End of Treatment) of Inflammation (Erythema) Evaluated by Mexameter of the Target Area as Compared to the Control Area at End of Follow-up
Description: Higher values describe a higher level of erythema.
Time Frame: week 6
Measure: Mean (Standard Deviation); unit: arbitrary units
Arm/Group | Blue Light | Control
Number analyzed (Participants) | 20 | 20
arbitrary units | -3.6 (9.38) | 1.2 (8.04)

5. Secondary Outcome: Change From Baseline of Patient Rating of Itching of the Target Area as Compared to the Control Area
Description: patients were asked to rate itching on a VAS scale (1 no itching; 100 worst imaginable itching)
Time Frame: week 4, 6
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Blue Light | Control
Number analyzed (Participants) | 20 | 20
units on a scale
  week 4 | -2.6 (20.72) | -15.6 (23.85)
  week 6 | -10.3 (26.25) | -19.6 (27.77)

6. Secondary Outcome: Change From Week 4 (End of Treatment) of Patient Rating of Itching of the Target Area as Compared to the Control Area at End of Follow-up
Description: patients were asked to rate itching on a VAS scale (1 no itching; 100 worst imaginable itching).
Time Frame: week 6
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Blue Light | Control
Number analyzed (Participants) | 20 | 20
units on a scale | -7.7 (14.11) | -4.0 (14.31)

7. Other Pre Specified Outcome: Hyperpigmentation - Evaluation by Mexameter
Description: Higher values describe a higher level of pigmentation.
Time Frame: week 0, 2, 4, 6
Measure: Mean (Standard Deviation); unit: arbitrary units
Arm/Group | Blue Light | Control
Number analyzed (Participants) | 20 | 20
arbitrary units
  week 0 | 27.8 (6.85) | 28.0 (7.99)
  week 2 | 26.3 (6.01) | 28.4 (6.04)
  week 4 | 25.6 (5.39) | 28.4 (7.71)
  week 6 | 26.5 (6.57) | 26.8 (5.51)

8. Other Pre Specified Outcome: Adverse Events (Serious and Non-serious)
Time Frame: week 0, 2, 4, 6
Measure: Number; unit: participants
Arm/Group | Blue Light | Control
Number analyzed (Participants) | 20 | 20
participants
  week 0 | 0 | 0
  week 2 | 0 | 0
  week 4 | 0 | 0
  week 6 | 0 | 0

9. Other Pre Specified Outcome: Adverse Device Events (Serious and Non-serious)
Time Frame: over 6 weeks
Measure: Number; unit: participants
Arm/Group | Blue Light | Control
Number analyzed (Participants) | 20 | 20
participants | 0 | 0

10. Other Pre Specified Outcome: Device Deficiencies
Description: This measure describes device deficiencies in general leading to a non functional device. No specific characteristics were assessed.
Time Frame: over 6 weeks
Measure: Number; unit: participants
Arm/Group | Blue Light | Control
Number analyzed (Participants) | 20 | 20
participants | 0 | 0

11. Other Pre Specified Outcome: Recovery of Hyperpigmentation During Follow up Period (Compared to Last Treatment)
Description: Higher values describe a higher level of pigmentation.
Time Frame: week 6
Measure: Mean (Standard Deviation); unit: arbitrary units
Arm/Group | Blue Light | Control
Number analyzed (Participants) | 20 | 20
arbitrary units | 0.9 (5.78) | -1.7 (6.49)

12. Other Pre Specified Outcome: Number of Participants With Acceptance of Hyperpigmentation at Week 6
Description: Questionaire if hyperpigmentation was acceptable if reported. Outcome was number of patients answering "yes" or "no".
Time Frame: week 6
Population: 7 patients out of 20 patients reported hyperpigmentation at week 6.
Measure: Number; unit: participants
Arm/Group | Blue Light
Number analyzed (Participants) | 7
participants
  Yes | 6
  No | 1

ADVERSE EVENTS:
Time Frame: Adverse events were collected throughout the whole study period after the patients signed the informed consent untill the last follow up visit (week 0 to week 6)
Arm/Group | Blue Light vs Control
Serious Adverse Events (participants affected / at risk) | 0/20
Other Adverse Events (participants affected / at risk) | 0/20

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No